CLINICAL TRIAL: NCT00352846
Title: Effect of Zoledronic Acid on Chemotherapy Induced Bone Loss in Non-Hodgkin's Lymphoma Patients Receiving Chemotherapy
Brief Title: Effect of Zoledronic Acid on Chemotherapy Induced Bone Loss
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2005-0698
Record Dates: First submitted 2006-07-13; First posted 2006-07-17 (Estimated); Results first posted 2013-06-20 (Estimated); Last update posted 2013-07-02 (Estimated); Status verified 2013-06

CONDITIONS: Non-Hodgkin's Lymphoma; Lymphoma
Keywords: Non-Hodgkin's Lymphoma; Lymphoma; Zoledronic Acid; Zoledronate; Zometa; Vitamin D; Calcium Carbonate; Bone Loss
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Lymphoma; Bone Diseases, Metabolic | interventions — Zoledronic Acid; Vitamin D; Calcium Carbonate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vitamin D + Calcium Carbonate (Experimental): Oral Vitamin D 400 mg daily + Calcium 1200 mg daily
  Interventions: Drug: Vitamin D; Drug: Calcium Carbonate
- Vitamin D + Calcium Carbonate + Zoledronic Acid (Experimental): Oral Vitamin D 400 mg daily and Calcium 1200 mg daily; Zoledronic Acid 4 mg/m^2 intravenous at baseline and 6 months.
  Interventions: Drug: Zoledronic Acid; Drug: Vitamin D; Drug: Calcium Carbonate

INTERVENTIONS:
Drug: Zoledronic Acid — 4 mg/m^2 by vein over 30 Minutes at baseline and 6 months.
  Other Names: Zometa; Zoledronate
  Arms: Vitamin D + Calcium Carbonate + Zoledronic Acid
Drug: Vitamin D — 400 mg by mouth daily
Drug: Calcium Carbonate — 1200 mg by mouth daily

SUMMARY:
Primary Objective:

* Evaluate the effect of zoledronate on change in bone mineral density (BMD) at the total lumbar spine and femoral neck.

Secondary Objectives:

* Evaluate the effect of zoledronate on change in BMD at the total hip
* Evaluate risk factors for developing osteoporosis on chemotherapy
* Determine correlative markers for response to zoledronate 4. Evaluate zoledronate effect on new bone fractures 5. Evaluate the cost-effectiveness of zoledronic acid (with calcium and vitamin D) versus standard treatment (calcium and vitamin D alone).

DETAILED DESCRIPTION:
Medicines called "bisphosphonates" have been shown to help people with cancer that has spread to their bones. Zoledronic acid is a "bisphosphonate". Some bisphosphonates are pills that can be swallowed. Other bisphosphonates such as zoledronic acid need to be given by vein (or intravenously). Some studies have shown that people with multiple myeloma, breast cancer, and prostate cancer that had spread to the bone had less side effects from their bone disease when they were treated with bisphosphonates by vein.

If you are found to be eligible to take part in this study, you will be randomly assigned (as in the toss of a coin) to one of two treatment groups. Participants in one group will receive standard care with calcium and Vitamin D alone. Participants in the other group will receive standard care with calcium and Vitamin D plus zoledronic acid. There is an equal chance of being assigned to either group. Both you and your study doctor will know if you are being treated with zoledronic acid.

You will be asked to come to the doctor's clinic 5 times over about 12 months (at the start of the study [baseline] and then every 3 months). Each visit should take about 1 hour. Participants in the zoledronic acid group will receive an infusion of zoledronic acid by vein at baseline and at 6 months into the study. The infusion will last about 30 minutes. This infusion procedure may or may not be done at the same time as your already scheduled chemotherapy treatment.

You will take calcium and Vitamin D pills while on study at amounts recommended for prevention of osteoporosis.

You will have a physical exam done at every visit. Various x-rays and/or bone density scans will be repeated after 12 months. Your doctor may also want to do additional bone density or x-ray scans if you have new symptoms or your symptoms get worse.

Before each treatment, you will have a blood test (about 1-2 teaspoons of blood) to make sure your kidneys are okay before each treatment with zoledronic acid. At each visit. your doctor or nurse will ask you how you are feeling and will ask about any medications you are taking or any medical problems you have had since your last visit. You will be asked to complete questionnaires about how you are feeling at certain visits. These questionnaires are 1 page long and should only take a few minutes to complete.

It is anticipated that your participation in this study will be 12 months. If your cancer gets worse, or if your doctor feels that you should be treated with a different medicine, you will be taken off of this study and your doctor will talk to you about other medicines that may be better for you.

Participants who received Zoledronic Acid will be contacted regularly to ask about any experience of osteonecrosis (bone death), for 10 years from the time they enroll on study. They will be interviewed by telephone call every 6 months.

This is an investigational study. Zoledronic acid is approved by the FDA for the treatment of high calcium levels in the blood. Zoledronic acid has not been approved by the FDA for what it is being used for in this study. After the treatment ends, you may continue to receive zoledronic acid or a similar drug, if your cancer doctor feels that it would help you. About 72 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of Non-Hodgkin's Lymphoma (B- or T-cell) or Hodgkin's lymphoma.
2. Prior Chemotherapy</= 4 weeks of treatment.
3. Age >/= 18 years old.
4. Eastern Cooperative Oncology Group (ECOG) Performance Status 0-3.
5. Estimated creatinine clearance >/= 60 ml/min.
6. Must sign an informed consent form.

Exclusion Criteria:

1. Radiologic evidence of vertebral or hip fracture.
2. BMD T-score less than (i.e., worse than or more negative than) -2.0 at any of the following sites: lumbar spine, femoral neck, or total hip.
3. Patients with secondary non-lymphomatous cancers metastatic to bone. However, other secondary cancers are allowed.
4. Spinal cord compression due to vertebral collapse.
5. Bisphosphonate treatment in the prior 6 months or steroid use (greater than 35 mg of prednisone equivalent steroids) in the prior 3 months. The use of topical, inhaled, or nasal steroids is allowed.
6. Primary hyperparathyroidism.
7. Active osteomalacia.
8. Untreated hypocalcemia (ionized, iCa), Ionized Ca level must be within normal limits prior to enrollment.
9. Untreated secondary hyperparathyroidism, Patients with abnormal parathyroid hormone (PTH) levels may be enrolled as long as they are being treated.
10. Untreated vitamin D deficiency, Vitamin D level may be abnormal and patient may be enrolled as long as they are being treated.
11. Untreated low testosterone (test in men only), testosterone level may be abnormal and patient may be enrolled as long as they are being treated.
12. Paget's disease.
13. Pregnant or breast-feeding.
14. Radiotherapy involving the mandible.
15. Current active dental problems including infection of the teeth or jawbone (maxilla or mandibular); dental or fixture trauma, or a current or prior diagnosis of osteonecrosis of the jaw (ONJ), or of exposed bone in the mouth, or of slow healing after dental procedures.
16. Recent (within 3 weeks) or planned dental or jaw surgery (e.g.. extraction, implants).
17. Patients with abnormal renal function as evidenced by either a serum creatinine greater than 3 mg/dL or by a calculated creatinine clearance of < 60 mL/minute.
18. Known hypersensitivity to zoledronic acid or other bisphosphonates.
19. Hypercalcemia: corrected Ca > 10.2 mg/dL or ionized Ca > 1.32 mmol/L

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2006-01; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fredrick Hagemeister, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Westin JR, Thompson MA, Cataldo VD, Fayad LE, Fowler N, Fanale MA, Neelapu S, Samaniego F, Romaguera J, Shah J, McLaughlin P, Pro B, Kwak LW, Sanjorjo P, Murphy WA, Jimenez C, Toth B, Dong W, Hagemeister FB. Zoledronic acid for prevention of bone loss in patients receiving primary therapy for lymphomas: a prospective, randomized controlled phase III trial. Clin Lymphoma Myeloma Leuk. 2013 Apr;13(2):99-105. doi: 10.1016/j.clml.2012.11.002. Epub 2012 Dec 29. PMID 23276888
- See also: MD Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: 01/27/2006 to 08/13/2009. All recruitments done at UT MD Anderson Cancer Center.
Pre-assignment Details: Of 135 enrolled participants, 61 were excluded from the trial before assignment to groups due to screen failures.
Period: Overall Study
Arm/Group | Vitamin D + Calcium Carbonate | Vitamin D + Calcium Carbonate + Zoledronic Acid
Started | 37 | 37
Completed | 29 | 24
Not Completed | 8 | 13
Not completed — Disease progression | 0 | 2
Not completed — Withdrawal by Subject | 3 | 8
Not completed — Ineligible | 3 | 2
Not completed — Non-compliance | 2 | 0
Not completed — Death | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vitamin D + Calcium Carbonate | Vitamin D + Calcium Carbonate + Zoledronic Acid | Total
Number analyzed (Participants) | 37 | 37 | 74
Age Continuous [Median (Full Range); unit: years] | 57 [19 to 75] | 61 [24 to 80] | 57 [19 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 14 | 27
  Male | 24 | 23 | 47
Region of Enrollment [Number; unit: participants]
  United States | 37 | 37 | 74

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change in Bone Mineral Density (BMD) T-Score From Baseline to 12 Months
Description: The 12-month change from baseline in BMD at the total lumbar spine. BMD evaluation was performed at baseline and at 12 months after initiation of therapy at the lumbar spine. BMD was measured by dual-energy, x-ray absorptiometry scanners. T-Score is the number of standard deviations above or below the mean. A T-score >= -1 indicates a normal BMD, while T-scores between -1 and -2.5 indicate osteopenia and T-scores <= -2.5 indicate osteoporosis.
Time Frame: From baseline to 12 Months
Population: BMD data available on 53 evaluable participants upon treatment completion.
Measure: Mean (Standard Deviation); unit: Percentage Change of BMD
Arm/Group | Vitamin D + Calcium Carbonate | Vitamin D + Calcium Carbonate + Zoledronic Acid
Number analyzed (Participants) | 29 | 24
Percentage Change of BMD | 0.08 (0.34) | -0.09 (1.23)

ADVERSE EVENTS:
Time Frame: 4 years, 3 months
Arm/Group | Vitamin D + Calcium Carbonate | Vitamin D + Calcium Carbonate + Zoledronic Acid
Serious Adverse Events (participants affected / at risk) | 0/37 | 0/37
Other Adverse Events (participants affected / at risk) | 0/37 | 0/37

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No